CLINICAL TRIAL: NCT03660683
Title: Cardio-Protective of Effect of Saxagliptin and Dapagliflozin Combination on Endothelial Progenitor Cells in Patients With Type 2 Diabetes
Brief Title: Effect of Saxagliptin and Dapagliflozin on Endothelial Progenitor Cell in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor did not want to continue funding the study
Sponsor: Sabyasachi Sen (Other)
Responsible Party: Sponsor-Investigator, Sabyasachi Sen, Associate Professor, Dept. of Medicine (Division of Endocrinology), George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180295
Record Dates: First submitted 2018-08-17; First posted 2018-09-06 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: saxagliptin dapagliflozin diabetes cardiovascular diseases EPC
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A Dapa (Experimental): Dapagliflozin 10 mg + Saxagliptin Placebo
  Interventions: Drug: Dapagliflozin 10mg
- Group B DapaSaxa (Active Comparator): Dapagliflozin 10mg + Saxagliptin 5mg
  Interventions: Drug: Dapagliflozin 10mg; Drug: Saxagliptin 5mg
- Placebo (Placebo Comparator): Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10mg PO QD
  Other Names: Farxiga
  Arms: Group A Dapa; Group B DapaSaxa
Drug: Saxagliptin 5mg — Saxagliptin 5 mg PO QD
  Other Names: Onglyza
  Arms: Group B DapaSaxa
Drug: Placebo Oral Tablet — Matching Placebo Tablets
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The Investigator hypothesize that Dapagliflozin will improve EPC number and function AND Saxagliptin in addition to Dapagliflozin (additive effect) may improve EPC number and function even more than Dapa alone, compared to placebo.

The Investigator propose a 3-arm randomized, parallel group, longitudinal study of 16-week intervention duration. Participants will be randomized to 3 groups:

Group A: Dapa (10 mg) + Saxa Placebo, Enroll n=15, retain n=12 Group B: Dapa (10 mg) + Saxa (5 mg), Enroll n=15, retain n=12 Group C: Dapa Placebo + Saxa Placebo, Enroll n=15, retain n=12

DETAILED DESCRIPTION:
The Investigator hypothesize that Dapagliflozin will improve EPC number and function AND Saxagliptin in addition to Dapagliflozin may have an additive effect to improve EPC number and function even more than Dapa alone, compared to placebo.

In this proposal the investigator plan to conduct a placebo matched study with type 2 diabetes subjects on any doses of metformin or Insulin or a combination of both and has no history of DPP4 ( Dipeptidyl Peptidase-4) DPP4 inhibitor, incretin mimetic or SGLT2 inhibitor intake history. Participants will have known macrovascular complications (such as Cardiovascular Disease (CVD), Cerebrovascular Accident (CVA), and Peripheral Vascular Disease (PVD).

3 STUDY OBJECTIVES

PRIMARY OBJECTIVE:

CELLULAR BIOMARKER OF ENDOTHELIUM

The primary objective is to ascertain if 16 weeks of Dapa or Dapa+Saxa Combo therapy will improve :

CD34+ cell number, CD34+ migratory function and CD34+ gene expression in type 2 diabetes with CVD.

SECONDARY OBJECTIVE:

ARTERIAL STIFFNESS AND RENAL FUNCTION, NON-CELLULAR MARKERS OF ENDOTHELIUM To determine whether use of Dapa or Dapa+Saxa Combo alters markers of endothelial function such as: arterial stiffness measures (via tonometry), biochemical measures derived from plasma, pertaining to endothelial function (hs-CRP, IL-6, TNF-alpha), renal function such as proteinuria (microalbumin/creatinine ratio) and urine exosome study to determine podocyte health. The secondary measures are indirect measures of endothelial inflammation in early type 2 diabetes patients.

Effect on Arterial Stiffness:

I. Pulse Wave Analysis and Vascular Flow will be assessed using SphygmoCor CP system from ATCOR as a measure of central arterial pressure and arterial stiffness.

II. Vessel health will be assessed by degree of arterial stiffness, using arterial tonometry.

III. The central and the aortic pressure is assessed by pulse wave analysis (PWA) and pulse wave velocity (PWV).

Effect on Blood Biochemistry:

The Investigator believes cell based biomarkers are superior to traditional serum and plasma biomarkers and the outcome report will be stronger if one can show positive correlation between the two outcome measures. The Investigator therefore will be looking at:

I. Inflammation, apoptosis and anti-oxidant protein levels: Highly selective C-reactive protein (hs-CRP), IL-6, TNF-alpha.

II. Plasma SDF1 alpha (ELISA) and GLP-1 and Ghrelin (ELISA) will be estimated to assess endothelial health and factors that may influence CD34+ cell chemotaxis III. Podocyte health via urine exosome analysis. IV. The glomerular filtration rate (GFR) will be estimated by MDRD equation.

a. GFR = 141 X min (Scr/κ,1)α X max(Scr/κ,1)-1.209 X 0.993Age X 1.018 [if female] X 1.159 [if African American]; where Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.32

TERTIARY OBJECTIVE:

METABOLISM MARKERS The tertiary objective is to determine whether use of Dapa or Dapa+Saxa Combo alters body composition, fasting lipid profile, and levels of insulin, glucose, and appetite controlling hormones.

Effect on Blood Biochemistry:

The Investigator believes cell based biomarkers are superior to traditional serum and plasma biomarkers and the outcome report will be stronger if one can show positive co-relation between the two outcome measures.

I. Fasting glucose, and insulin. a. Glycemic control will be evaluated by measuring fasting blood glucose, insulin levels and HbA1c. Fasting blood glucose, insulin and lipid profile will be used to assess insulin resistance.28,31 II. Lipid profile III. Appetite controlling hormones via LabCorp: Leptin, Adiponectin IV. Appetite controlling hormones, via ELISA: GLP1, Ghrelin

Effect of Dapa and Dapa+Saxa Combo on Body Habitus (Determination of body composition and visceral fat) The Investigator plans to study cardio-metabolic effect of Dapa and Dapa+Saxa Combo.

I. Using body composition scale:

1. Height and weight will be measured and the body mass index (BMI=kgm2) used as an indicator of relative weight.
2. The body composition scale calculates body fat%, total body water%, fat free mass, etc., in addition to BMI.

   The secondary outcome markers (arterial stiffness and renal outcome measures) and tertiary outcome markers (serum biochemistry) are crucial in order to corroborate the cellular findings with currently accepted clinical efficacy outcome measures such as arterial stiffness and serum biochemistry. This design is similar to our recently published manuscript on Saxagliptin and cellular outcome measures.

   4 INVESTIGATIONAL PLAN

   STUDY DESIGN AND DURATION

   +/- 6 day window for visits

   *Assessed at week 0, 8 and 16: Primary, Secondary & Tertiary Outcomes.

   Week 20: A telephone call to subjects will be made 4 weeks after last dose of study medication to determine if there have been any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study, and provide a signed & dated informed consent.
2. Diagnosis of Type 2 diabetes mellitus using criteria of the American Diabetes Association.
3. 30-70 years old.
4. HbA1C 7 to 10%, both inclusive
5. BMI of 25 - 39.9 kg/m2 both inclusive.
6. Taking a stable dose (for 12 weeks) of Metformin (any dosage) and/or Insulin (any dosage) for the treatment of T2DM
7. Patients with current Cardiovascular Disease (CVD) in tye 2 diabetes patients, defined by ≥ 1 of the following:

   1. MI >2 months prior
   2. Multivessel CAD
   3. Angina (intermittent or chronic)
   4. Single vessel CAD with positive stress test or UA hospitalization in prior year
   5. UA >2 months prior and evidence of CAD
   6. Stroke >2 months prior
   7. Occlusive PAD
   8. Proteinuria of more than 30mg/dl

Exclusion Criteria:

1. Planned CV surgery or angioplasty in 1 month
2. Prior surgery with chronic malabsorption (eg, bariatric) in prior 1 year
3. Diagnosis of Type 1 diabetes mellitus
4. History of GAD antibody positive status
5. Uncontrolled Inflammatory Disease/Inflammatory drug use. **Evaluated by PI on case-by-case basis**
6. Recent history of diabetic keto-acidosis in the past 3months, or recurrent history of diabetic ketoacidosis (≥ 3 times)
7. Active bladder cancer
8. Active wounds (e.g. Diabetic ulcers) or recent surgery within 1 month
9. Untreated hyper/hypothyroidism
10. Women of child bearing potential who are not willing to use a contraceptive method to avoid pregnancy for the 16 weeks of study duration
11. Women who are pregnant or breastfeeding
12. Implanted devices (eg. Pacemaker) that may interact with Tanita scale
13. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial Concomitant Medications
14. Taking any other oral anti-diabetic agent other than Metformin and/or Insulin for their treatment of T2DM
15. Beginning statin medications in the past 1 month or change in statin dose in the past 1 month
16. Use of consistent long-term steroid medication (oral, inhaled, injected) within the last 1 month
17. Treatment with a strong cytochrome P450 3A4 (CYP34A) or P-gp inducer (ie. Rifampin)
18. Subjects with a history of any serious hypersensitivity reaction to Dapagliflozin / Saxagliptin or another SGLT-2 inhibitor/ DPP4 inhibitor Laboratory Findings
19. Uncontrolled hyperglycemia, defined as a fasting glucose >240 mg/dL (>13.3 mmol/L) at screening.
20. Liver disease with ALT, AST or ALP x3 ULN
21. eGFR < 60 mL/min/1.73 m2 by MDRD equation in the past 3 months
22. Clinically significant RBC disorders such as hemoglobinopathies
23. Serum creatinine levels ≥1.8 mg/dL with estimated eGFP < 60 mL/min
24. Triglycerides > 450 mg/dL
25. Baseline Hematuria (judged by a urinalysis dipstick at screening) Social History
26. Active smokers
27. Chronic or persistent alcohol or drug abuse
28. Prisoners or subjects who are involuntarily incarcerated
29. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg. infectious disease) illness
30. Participation in another trial with an investigational drug within 30 days prior to informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, PhD, Principal Investigator — GWU
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nandula SR, Jain A, Sen S. Cardio-renal effect of dapagliflozin and dapagliflozin- saxagliptin combination on CD34 + ve hematopoietic stem cells (HSCs) and podocyte specific markers in type 2 diabetes (T2DM) subjects: a randomized trial. Stem Cell Res Ther. 2025 Jan 26;16(1):28. doi: 10.1186/s13287-025-04130-x. PMID 39865301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Started | 4 | 5 | 6
Completed | 4 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 11
  >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 5 | 6
  Male | 4 | 4 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 4 | 8
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 104 (5.7) | 125 (9.9) | 138.8 (18.0) | 127.4 (18.1)
  Diastolic | 69.5 (0.7) | 78 (2.4) | 82.5 (13.5) | 78.8 (10.3)
CD34+ Cell Fraction [Mean (Standard Deviation); unit: percentage of WBC] — Quantifying CD34+ cells is based on proportion of the monocytes that are CD34+ to account for any variations in cell harvesting or death during analysis.
  percentage of WBC | 0.61 (0.77) | 2.35 (1.79) | 3.55 (1.74) | 2.23 (1.78)
Colony Forming Units (Day 14) [Mean (Standard Deviation); unit: cfu (integer)] | 18.9 (26.9) | 12.6 (6.9) | 9.7 (7.6) | 13.4 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: CD 34+ Cell Migratory Function
Description: Proportion of cells that migrate through SDF1a in a transwell assay. This proportion is represented as a migratory rating scale from 0-1, with 1 being 100% of cells migrate. A larger value indicates better migratory function of the CD34+ cells.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
score on a scale | 0.675 (0.094) | 0.75 (0.096) | 0.253 (0.352)

2. Secondary Outcome: CD 34+ Cell Gene Expression
Description: Fold change of Gene Expression in T2Dm with CVD relative to visit 1
Time Frame: 16 weeks from visit 1
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
fold change
  CAT | 2.57 (0.52) | 7.12 (2.14) | 1.71 (0.28)
  CXCL12 | 6.83 (2.87) | 4.23 (0) | 2.34 (0.44)
  CXCR4 | 1.71 (0.27) | 0.56 (0.07) | 1.08 (0.08)
  EDN1 | 2.67 (0.79) | 0.89 (0.06) | 0.82 (0.08)
  GAPDH | 2.87 (0.56) | 3.22 (0.86) | 4.23 (1.05)
  GPX3 | 0.89 (0.14) | 0.65 (0.09) | 3.37 (0.29)
  IL6 | 1.08 (0.18) | 0.17 (0.02) | 2.97 (0.48)
  KDR | 0.70 (0.13) | 0.44 (0) | 1.76 (0.26)
  NOS3 | 1.63 (0.40) | 4.16 (0.88) | 0.99 (0.11)
  P21 | 1.11 (0.16) | 1.55 (0.27) | 1.23 (0.04)
  PECAM1 | 2.86 (0.39) | 6.19 (1.21) | 1.69 (0.14)
  SOD2 | 1.96 (0.23) | 2.23 (0.41) | 2.19 (0.37)
  TNF | 1.76 (0.22) | 0.79 (0.14) | 1.12 (0.10)
  TP53 | 2.41 (0.63) | 3.53 (1.07) | 1.55 (0.21)
  VEGFA | 1.41 (0.19) | 6.14 (2.05) | 1.29 (0.13)

3. Secondary Outcome: CD 34+ Cell Fraction
Description: Quantifying CD34+ cells is based on proportion of the monocytes that are CD34+ to account for any variations in cell harvesting or death during analysis.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
percentage of cells | 1.15 (0.33) | 3.17 (0.27) | 1.74 (0.31)

4. Secondary Outcome: Arterial Stiffness - Augmentation Index
Description: Augmentation index was calculated via tonometry with Sphygmocor Device (Pulse Wave Analysis). Augmentation index is calculated as the augmentation pressure (the amplitude of the reflected pulse wave) divided by the pulse pressure (systolic - diastolic) * 100 to give a percentage of pulse pressure. The software then calculates an estimated Augmentation Index at heart rate of 75 as a form of "normalization." Lower values are generally preferred as they indicate more pliable and healthy arteries.
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: percentage of pulse pressure
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
percentage of pulse pressure
  Aug Index | 13.67 (2.17) | 34 (2.83) | 25.65 (0.15)
  Aug Index @75 Heart Rate | 12 (1) | 30 (3.96) | 27.75 (1.0)

5. Secondary Outcome: Blood Biochemistries
Description: hsCRP
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mg/L | 1.265 (0.975) | 1.408 (1.106) | 4.258 (1.799)

6. Secondary Outcome: Renal Function
Description: Microalbumin/Creatinine Ratio (Proteinuria)
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: mcg/mg
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mcg/mg | 37.3 (11.9) | 13.22 (0.96) | 158.48 (47.76)

7. Secondary Outcome: Urine Exosome Assay
Description: Protein western analysis of Exosomes released from Kidney Podocyte is a indicator of kidney Podocyte health.
  Expressed as a ratio normalized to CD9 expression
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
ratio
  Nephrin | 1.16 (0.10) | 0.49 (0.10) | 0.67 (0.13)
  Podocalyxin | 2.59 (0.43) | 2.10 (0.48) | 0.79 (0.01)

8. Secondary Outcome: Arterial Stiffness
Description: Pulse Wave Velocity
Time Frame: Week 16
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
m/s | 8.23 (0.16) | 8.1 (0.14) | 9.55 (0.22)

9. Secondary Outcome: Arterial Stiffness - Augmentation Pressure
Description: Augmentation index was calculated via tonometry with Sphygmocor Device (Pulse Wave Analysis). Augmentation index is calculated as the augmentation pressure (the amplitude of the reflected pulse wave) divided by the pulse pressure (systolic - diastolic) * 100 to give a percentage of pulse pressure. The software then calculates an estimated Augmentation Index at heart rate of 75 as a form of "normalization." Lower values are generally preferred as they indicate more pliable and healthy arteries.
  Here, augmentation pressure is shown as a reference for the Augmentation Index calculations in the previous section.
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mmHg | 4.0 (0.66) | 13.5 (1.55) | 6.77 (0.77)

10. Other Pre Specified Outcome: Fasting Lipid Profile
Description: Total Cholesterol, LDL, HDL and VLDL
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mg/dL
  Total Cholesterol | 155.5 (7.2) | 119.8 (3.1) | 149.4 (5.6)
  HDL | 41.5 (1.2) | 37.8 (2.5) | 40.8 (1.4)
  VLDL | 20.0 (1.4) | 30.8 (4.4) | 25.4 (2.5)
  LDL | 94.0 (0.7) | 51.2 (3.1) | 83.2 (4.0)

11. Other Pre Specified Outcome: Serum Insulin Level
Description: Measured in fasting state at visit
Time Frame: 16 Weeks
Measure: Mean (Standard Error); unit: mcU/mL
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mcU/mL | 15.5 (2.3) | 15.8 (1.9) | 20.2 (2.7)

12. Other Pre Specified Outcome: Serum Glucose
Description: Fasting Glucose level measured in serum
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
mg/dL | 113.5 (13.5) | 106.4 (24.3) | 184.8 (41.6)

13. Other Pre Specified Outcome: Appetite Controlling Hormone
Description: Leptin, (Adiponectin, GLP1, Ghrelin in separate entry)
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
ng/mL | 8.13 (3.83) | 25.60 (15.64) | 80.96 (55.56)

14. Other Pre Specified Outcome: Serum Glucose
Description: HbA1C (estimate of serum glucose over 3 months)
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
Number analyzed (Participants) | 4 | 5 | 6
percentage of hemoglobin | 8.53 (3.16) | 2.43 (1.62) | 8.80 (1.47)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from signing of informed consent until 30 days after the last patient visit (approximately 20 weeks(
Arm/Group | Group A Dapa | Group B DapaSaxa | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
Study is limited by the small cohort used in each group. Many visit 2 data points missing, reported analysis only performed with visit 1 and 3 data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT03660683/Prot_SAP_000.pdf